CLINICAL TRIAL: NCT02268422
Title: A Two-period, Randomised, Open-label, Crossover, Pharmacokinetic Study to Assess the Bioequivalence and Adhesion of Buprenorphine Transdermal System Second Generation Patch Compared With First Generation Patch, in Healthy Volunteers
Brief Title: Bioequivalence and Adhesion Comparison of Buprenorphine Patches
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BUP1507; 2014-002116-17 (EudraCT Number)
Record Dates: First submitted 2014-10-09; First posted 2014-10-20 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Pain
Keywords: Healthy volunteer; crossover; open-label; randomised; bioequivalence; pharmacokinetic study
MeSH Terms: conditions — Pain | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7 day patch (Experimental): Buprenorphine transdermal system (BTDS) 2nd generation
  Interventions: Drug: Buprenorphine
- 7 Day Patch (Active Comparator): 1st Generation BTDS: Butrans
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — 7 day patch

SUMMARY:
To compare a 2nd generation Buprenorphine Transdermal System (BTDS) patch with a marketed 1st generation BTDS patch to confirm that the two are bioequivalent (deliver the same amount of drug) and that they equally both stick to the skin over 7 days of continuous wear.

DETAILED DESCRIPTION:
The objective is to compare a 2nd generation BTDS patch 20 µg/h to the 1st generation patch to confirm bioequivalence. Determination will be via measurement of drug concentrations in the blood at serial collection time points pre-dose until 288 hours post-patch application. Approximately 100 healthy male and female volunteers will receive both BTDS patches across two study periods with a 14-day wash-out between applications.

Each patch will be worn for 7 consecutive days and the study will also review the adhesion of each patch to the skin of the subjects. The overall safety and tolerability of both patches will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Healthy male or female subjects aged 18 to 55 inclusive.
3. Female subjects of child bearing potential must be willing to use two highly effective methods of contraception throughout the study, one of which must include a barrier method. A highly effective method of birth control is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, combined oral contraceptives, some IUDs (Intrauterine Device), true sexual abstinence when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence e.g. calendar, ovulation, symptothermal, post-ovulation methods, declaration of abstinence for the duration of the trial, and withdrawal are not acceptable methods of contraception) or vasectomised partner. Acceptable barrier methods are either their partner's use of a condom or the subject's use of an occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
4. Female subjects who are postmenopausal (defined as spontaneous amenorrhoea for at least 1 year) or permanently sterilised (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy). These subjects are not required to use any contraception.
5. Male subjects who are willing to use contraception with their partners throughout the study and for 30 days after completion of the study and agree to inform the Investigator if their partner becomes pregnant during this time.
6. Body weight ranging from 55 to 100 kg and a BMI ≥ 18.5 and ≤ 29.9.
7. Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, laboratory tests and ECG.
8. Willing to eat all the food supplied throughout the study.
9. The subject's primary care physician has confirmed within the last 12 months of the initial dosing date, that there is nothing in the subject's medical history that would preclude their enrolment into a clinical study.
10. Will refrain from strenuous exercise during the entire study. They will not begin a new exercise program nor participate in any unusually strenuous physical exertion.

Exclusion Criteria:

1. Female subjects who are pregnant or lactating.
2. Any history of drug or alcohol abuse.
3. Any history of conditions that might interfere with drug absorption, distribution, metabolism or excretion.
4. Use of opioid or opioid antagonist-containing medication in the past 30 days.
5. Any history of frequent nausea or vomiting regardless of aetiology.
6. Any history of seizures or symptomatic head trauma.
7. Participation in a clinical drug study during the 90 days preceding the initial dose in this study, or participation in any other clinical drug study during this study.
8. Any significant illness during the 4 weeks preceding entry into this study.
9. A history of additional risk factors for Torsades de Pointes (e.g. heart failure, hypokalaemia, personal or family history of long QT syndrome, syncope, or family history of sudden death).
10. Abnormal cardiac conditions including any of the following:

    * QTcF interval greater than 450 msec at screening or at check-in before first dosing.
    * Increase in QTcF of more than 60 msec above pre-dose values of each study period or QTcF > 500 msec at any time during the study.
11. Use of medication within 5 times the half-life or minimum 14 days for prescription medication or 7 days for over-the-counter preparations (including vitamins, herbal and/or mineral supplements), whichever is longer, before the first dose of study treatment and during the study (with the exception of the continued use of Hormone Replacement Therapy (HRT) and contraceptives). Note: subjects taking oral contraceptives containing CYP3A4 inhibitors such as gestodene should be excluded as this may lead to elevated plasma concentrations.
12. Refusal to abstain from caffeine or xanthine containing beverages and grapefruit juice within 48 hours before IMP administration until after the last study PK sample has been taken in each study period.
13. Weekly alcohol intake exceeding the equivalent of 14 units/week for females and 21 units/week for males.
14. Consumption of alcoholic beverages within 48 hours before IMP administration, and refusal to abstain from alcohol for the duration of the study confinement and for at least 48 hours after the last naltrexone dose in each study period.
15. History of smoking within 45 days of IMP administration and refusal to abstain from smoking during the study.
16. Blood or blood products donated within 90 days prior to IMP administration or any time during the study, except as required by this protocol.
17. Positive results of urine drug screen, alcohol test, pregnancy test, HBsAg, Hepatitis C antibody, or HIV tests.
18. Known sensitivity to buprenorphine, naltrexone, related compounds or any of the excipients or any contraindications as detailed in the Butrans Summary of Product Characteristics or Nemexin Summary of Product Characteristics.
19. Clinically significant history of allergic reaction to wound dressings or elastoplast.
20. Subjects with any dermatological disorder or tattoos at the proposed sites of patch application, or with a history of eczema/cutaneous atrophy.
21. Subjects who will not allow hair to be removed at the proposed patch application sites which may prevent proper placement of the patch.
22. Refusal to allow their primary care physician to be informed of participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Up to 288 hours
  Pharmacokinetics parameters AUC and Cmax assessments
Patch adhesion | 168 hours
  Patch site adhesion

SECONDARY OUTCOMES:
Residual Buprenorphine content following 7 days of wear | 168 hours
  Determination of residual Buprenorphine content remaining in both BTDS patches following removal
Measure of Safety and tolerability | From screening to 40 days after patch application
  Adverse event assessment from all subjects over the entire study

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Croydon
  - Nottingham